CLINICAL TRIAL: NCT03731104
Title: Changes in Cerebral Circulation and Oxygenation During Hemodynamic Resuscitation in Critically Ill Children Without Head Trauma
Brief Title: Cerebral Circulation in Critically Ill Children
Acronym: CIRCU-REAPED
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A01392-53
Record Dates: First submitted 2018-08-17; First posted 2018-11-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Arterial Hypotension; Shock; Cerebral Lesion
Keywords: Near InfraRed Spectroscopy; Brain perfusion; Pediatric shock; Catecholamines
MeSH Terms: conditions — Hypotension; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Near InfraRed Spectroscopy assessment — Regional Cerebral Oxygen saturation (rScO2 ) values will be collected for all patients during the procedure using a 2-wavelength (730-810 nm) cerebral oxymeter (monitor INVOS 5100C®, Medtronics). Two transducers will be placed on both fronto-parietal sides of the patient's head.
  To assess the balance between oxygen delivery and consumption, the Fractional cerebral Tissue Oxygen Extraction (FTOE) will be calculated as this ratio: FTOE=[SpO2-rScO2]/SpO2.
  Data will be collected for a period of 3 hours starting from the beginning of catecholamine treatment.
  Other Names: NIRS assessment
Device: Transcranial Doppler Ultrasound assessment — Transcranial Doppler ultrasound will be performed for all patients during the procedure using a VIVID S-5 (General Electric®) echograph. All examinations will be performed by a single trained operator. A 3 MHz probe will be placed on left and right temporal window to detect signal from the middle cerebral artery. 2 measures will be performed for each side to have the mean of the two measures; In case of difference in measures of more than 20%, a third measure will be performed.
  Measures will be performed for a period of 3 hours starting from the beginning of catecholamine treatment.
  Other Names: TCD assessment
Device: Cardiac output assessment — Transthoracic echocardiography will be realized for all patients during the procedure using a transthoracic ultrasound device (VIVID S-5, General Electric®) with a 3 to 6 MHz probe. All examinations will be performed by a single trained operator.
  Two echocardiographic views will be examined to assess cardiac output : the two-chamber long-axis view to measure sub-aortic diameter (d), and the four-chamber view to measure the Left ventricular outflow tract velocity time integral (LVOT VTI). Cardiac output (Qc) will then be calculated taking account these parameters and heart rate with this formula : Qc = [π x d2 x VTI x HR] / 4 2 measures will be performed to have the mean of the two measures; In case of difference in measures of more than 20%, a third measure will be performed.
  Measures will be performed for a period of 3 hours starting from the beginning of catecholamine treatment.

SUMMARY:
The principal purpose of this study is to describe the changes in cerebral circulation (assessed by transcranial ultrasound) and oxygenation (assessed by Near InfraRed spectroscopy, NIRS) during resuscitation for hemodynamic failure (arterial hypotension or shock) in critically ill children treated with vasoactive or inotropic drugs.

The secondary objectives are :

i) to evaluate the association between an alteration of cerebral circulation and/or oxygenation and an alteration in macro-circulatory parameters (Mean Arterial Blood Pressure and cardiac output) or a bad outcome, ii) to study if cerebral autoregulation is impaired

DETAILED DESCRIPTION:
Pediatric shock is a frequent and serious cause of hospitalization in pediatric intensive care unit that can lead to multi-organ failure and death.

Its early recognition improves patients' outcome, as well as the establishment of targeted guidelines pursuing normalization of macro-circulatory parameters (ie blood pressure and lactate).

However, regional hypoperfusion leading to organ failure can be present before the alteration of these parameters, and persist after their restoration.

Brain lesions are common in critically ill children with cerebral hypoperfusion, since they may have impaired autoregulation and permeable blood-brain barrier. Vasoactive and inotropic drugs used for hemodynamic resuscitation should restore systemic and regional circulation, but may be inadequate on brain perfusion because of i) their variable and unpredictable cardiovascular effects , and ii) a strong interindividual variability between patients. As such, the impact of this medication on cerebral circulation and oxygenation is unknown.

Monitoring cerebral circulation and oxygenation during a hemodynamic resuscitation using catecholamines is a first step to identify risk factors of an altered brain perfusion, and to improve treatment of shock.

ELIGIBILITY:
Inclusion Criteria:

Neonates and children from 0 to 18 years old hospitalized in pediatric intensive care unit (PICU) with hemodynamic failure requiring vasoactive or inotropic treatment. This includes :

* shock (tachycardia, troubles of peripheral perfusion with capillary refill time >3 sec, oliguria, with or without alteration of consciousness or arterial hypotension)
* isolated arterial hypotension if it needs medical treatment to readjust balance between oxygen demand and oxygen consumption

Exclusion Criteria:

* primitive cerebral lesion: traumatic or neurosurgical (including brain death states)
* preterm neonates of less than 37 weeks gestational age
* patients already receiving more than one catecholamine
* patients too instable, defined by a respiratory instability (pulse oxymetry of less than 80% during more than 5 minutes) and/or hemodynamic instability (variability of blood pressure and heart rate of more than 50%) and/or cardiorespiratory arrest.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients hospitalized in 4 french Pediatric Intensive Care Units
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Near InfraRed Spectroscopy (NIRS) | 3 hours
  rScO2 and FTOE variations (left and right). A cerebral desaturation will be defined by a rScO2 delta >20% from the baseline value (before premedication).
Variations of velocities of middle cerebral artery (left and right), in cm/s | 3 hours
  Transcranial Doppler ultrasound
Variations of pulsatility index of middle cerebral artery (left and right) | 3 hours
  Transcranial Doppler ultrasound
Variations of resistance index of middle cerebral artery (left and right) | 3 hours
  Transcranial Doppler ultrasound

SECONDARY OUTCOMES:
Mean arterial pressure | 3 hours
  Correlation between microcirculatory parameters (transcranial Doppler ultrasound and NIRS) and mean arterial pressure
Cardiac output calculated with Left ventricular outflow tract velocity time integral (LVOT VTI) measured by cardiac ultrasound | 3 hours
  Correlation between microcirculatory parameters (transcranial Doppler ultrasound and NIRS) and cardiac output (Qc), which will be calculated taking account these parameters and heart rate with this formula : Qc = [π x d2 x VTI x HR] / 4
PEdiatric logistic organ dysfunction score (PELOD-2) | 3 hours
  Correlation between cerebral perfusion (transcranial Doppler ultrasound and NIRS) and Organ Dysfunction assessed by PELOD-2 score.
  PELOD-2 score includes 10 variables corresponding to 5 organ dysfunctions. Values extend from 0 (best outcome) to 33 (worst outcome).
Death in pediatric intensive care unit | 3 hours
  Correlation between cerebral perfusion (transcranial doppler ultrasound and NIRS) and outcome (PELOD-2, death in PICU = pediatric intensive care unit)
Cerebral autoregulation evaluation | 3 hours
  Cerebral autoregulation will be estimated thanks to a Pearson coefficient correlation between mean arterial pressure (MAP) and rScO2. A ratio MAP/rScO2 > 0,5 defines an impaired cerebral autoregulation

CONTACTS AND LOCATIONS:
Overall Officials: Meryl VEDRENNE-CLOQUET, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Hôpital Trousseau, Paris
  - Hôpital Necker, Paris
  - Hôpital Robert Debré, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vedrenne-Cloquet M, Chareyre J, Leger PL, Genuini M, Renolleau S, Oualha M. Low Dosing Norepinephrine Effects on Cerebral Oxygenation and Perfusion During Pediatric Shock. Front Pediatr. 2022 Jul 6;10:898444. doi: 10.3389/fped.2022.898444. eCollection 2022. PMID 35874564